CLINICAL TRIAL: NCT04283864
Title: Decoding Personalized Nutritional, Microbiome and Host Patterns Impacting Clinical and Prognostic Features in Crohn's Disease
Status: Recruiting | Type: Observational
Sponsor: Weizmann Institute of Science (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Eran Elinav, Principal Investigator, Host-Microbiome Interaction Research Group, Weizmann Institute of Science
Other Study IDs: 0722-19 -RMC
Record Dates: First submitted 2019-11-19; First posted 2020-02-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; microbiome; Personal diet; personalized nutrition; Nutribiome
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A
- Group B
- Group C

SUMMARY:
The study is 3 arms observational study with no intervention that aims to understand the link between Crohn's disease, microbiome and diet in children.

150 children newly diagnosed with Crohn's disease will participate in the study and their data will be used to create an algorithm about their microbiome, disease, diet, etc.

100 other children newly diagnosed will participate in the study and their data will be use to validate the algorithm.

The investigators will be recruiting 50 healthy participants: 20 that are undergoing an endoscopy for abdominal pain and 30 that comes to the physician for different reasons.

After parental consent, the participants will receive an explanation of the study and sign a consent form for colonoscopy. Before colonoscopy, participants will bring fecal samples, give blood samples, biopsies and biopsy brushes (superficial scraping of the tissue) will be taken during the operation. These samples will be retained until further consent is obtained for further study.

After receiving the results of the colonoscopy, children who have been diagnosed with Crohn's disease will be offered to participate in the second part of the study, they will receive an explanation about the app, collection of fecal samples at home, diet logs and anthropometric measurements, demographic information, medical and family history will be registered.

During the first 3 months: the participants will be asked to log data in the app and collect fecal samples at home. They will be asked to come for a follow up visit where anthropomorphic measurements and blood samples will be taken.

Participants will be asked to log in every day to report in the app daily activity and food intake throughout the study period. Each week, the research coordinator will call on participants to make sure the app is correctly filled in, collect the stool samples correctly and answer questions. During the entire study participants will collect fecal samples, every first week of the month participants will enter information in the app.

For children who have not been diagnosed with Crohn's disease by the colonoscopy, or children who visit the institute for reasons other than inflammatory bowel disease without a clear finding will participate in the study control group. If consent is given, fecal samples will be collected at the entrance of the study and after one year, blood samples, a food questionnaire and anthropometric indices, demographic information, medical and family history will be completed.

ELIGIBILITY:
Inclusion Criteria:

* CD study group - 'Consent form - Part 1'

  1. Children with clinical suspicion for CD.
  2. Between 6 and 18 years of age.
  3. Naïve to any medical or nutritional intervention.

CD study group - 'Consent form - Part 2'

1. Children with CD confirmed by endoscopy (and based on accepted criteria7)
2. Between 6 and 18 years of age.
3. Naïve to any medical or nutritional intervention.

Control group undergoing endoscopy en between 6 and 18 years of age undergoing colonoscopy for non-specific abdominal pain or other non-inflammatory gastrointestinal conditions.

Control group not undergoing colonoscopy

1. Children with no symptoms or signs of gastrointestinal disease and no known medical conditions.
2. Children between 6 and 18 years of age. These children will be recruited from general pediatric clinics (children attending for routine check-up), orthopedic clinics, ophthalmology clinics or schools.

Exclusion Criteria:

* CD study group

  1. Chronic treatment with any drug upon enrolment and the use of systemic antibiotics, probiotics or proton pump inhibitors during 30 days prior to enrollment.
  2. Morbid obesity (BMI > 95th percentile for their age and gender).
  3. Following particular dietary regimen/dietitian consultation/participation in another study.
  4. Chronic use of steroids or immunomodulatory medications prior to CD diagnosis.
  5. Any other chronic disease (e.g. HIV, Cushing disease, acromegaly, hyperthyroidism, etc.), cancer and recent anti-cancer therapy, neuro-psychiatric disorders, coagulation disorders, celiac disease or any other chronic GI disorder.
  6. Gut-related surgery, including bariatric surgery.
  7. Inability of the participant and nuclear family to follow and utilize the smartphone application.

Control group not undergoing colonoscopy

1. Children with no symptoms or signs of gastrointestinal disease and no known medical conditions.
2. Children between 6 and 18 years of age. These children will be recruited from general pediatric clinics (children attending for routine check-up), orthopedic clinics, ophthalmology clinics or schools.

Control group undergoing endoscopy

1. Any known chronic illness.
2. Following particular dietary regimen/dietitian consultation/participation in another study.
3. Chronic treatment with any drug upon enrolment and the use of systemic antibiotics, probiotics or proton pump inhibitors during 30 days prior to enrollment.
4. Gut-related surgery, including bariatric surgery.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children between 6 to 18 years old. 250 with crohn disease ( undergoing endoscopy) 20 children without Crohn Disease ( undergoing endoscopy) 30 healthy children ( not undergoing endoscopy)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Personalised nutrition Algorithm based on microbiome. | 3 years
  Using machine learning we will create a trained personalised decision-tree based predictor enabling a significant prediction of nutritional impacts on CD clinical and inflammatory features during the first year of follow-up. It will be based on information gathered from microbiome ( metagenomic and 16s sequencing of stool microbiome), nutritional questionnaire and disease states (via fecal calprotectin test) in children with Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Eran Elinav, Prof, Principal Investigator — Weizmann Institute of Science
Locations (2):
- Schneider children's medical center, Petah Tikva, Israel
- University of Naples "Federico II", Naples, Italy

IPD SHARING:
Plan to Share IPD: No